CLINICAL TRIAL: NCT02081417
Title: Patient-Centered Trauma Treatment for PTSD and Substance Abuse: Is it an Effective Treatment Option?
Brief Title: Effectiveness of Peer-Delivered Trauma-Specific Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4484
Record Dates: First submitted 2014-03-03; First posted 2014-03-07 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Post-Traumatic Stress Disorder; Substance Use Disorders
Keywords: Trauma; Post traumatic stress disorder; substance use disorders; peer-delivered trauma treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer led (Other): Number sessions of the intervention of an evidenced based practice called "Seeking Safety" led by a Peer (6 sessions will be used to define treatment completion)
  Interventions: Behavioral: Seeking Safety
- Clinician led (Other): Number intervention groups of an evidence based practice called "Seeking Safety" led by a master's level Clinician (6 sessions will be used to define treatment completion).
  Interventions: Behavioral: Seeking Safety

INTERVENTIONS:
Behavioral: Seeking Safety — SS is a present-focused clinical intervention designed to target trauma/PTSD and SUDs.

SUMMARY:
Patient-Centered Trauma Treatment, i.e., treatment delivered by peers with lived-experience, has the potential to increase access to trauma treatment in underserved communities. This could positively impact the lives of millions of people as 70% of adults in the U.S have experienced a traumatic event and the consequences of trauma are devastating and far reaching, including chronic and comorbid physical and mental health problems. The most known consequences of trauma include post-traumatic stress disorder (PTSD) and substance use disorders (SUDs). Seeking Safety (SS) is the most effective evidenced-based treatment for co-occurring trauma, PTSD and SUDs. While no specific degree or experience level is required to conduct SS, all the evidence comes from studies using trained clinicians to implement the treatment, including social workers, psychologists, and psychiatrists. However, these research findings do not generalize to underserved communities that lack mental health professionals. Innovative approaches to treatment, such as peer-delivered services, are required to meet the demand for care in underserved areas. While the benefits of peer-delivered services have been well-documented in many areas, the value of peers in the provision of trauma-treatment is unknown. A theoretical basis supports the potential for peer-delivered trauma-treatment to be effective in addition to the strong therapist-patient bond, (i.e. therapeutic alliance (TA), which is an important predictor of treatment outcome and a typical result of peer-patient relationships.

Our research question is whether there is a difference between peer-led SS (PL-SS) groups and clinician-led SS (CL-SS) groups in improving the lives of people with trauma, PTSD and SUDs?

The investigators have three specific aims:

1. Determine the effectiveness of PL-SS groups compared to CL-SS groups in decreasing substance use and PTSD symptoms and improving coping skills, overall mental health and physical health. Hypothesis: PL-SS compared to CL-SS groups will be as effective in improving outcomes.
2. Compare levels of TA among PL-SS and CL-SS groups and examine the impact of TA on outcomes.Hypotheses: Levels of TA will be higher and will play more of a role in impacting outcomes in the PL-SS compared to CL-SS groups.
3. Determine if the standard Seeking Safety Instructor Training (SS-IT) is adequate for peers. Hypothesis: Peers will identify topics that will enhance the SS-IT.

ELIGIBILITY:
Inclusion Criteria:

* Be a member of INSIDE OUT, a peer-run wellness center
* Be at least 18 years old
* Have a history of trauma
* Meet DSM-IV diagnostic criteria for lifetime and current full or sub-threshold PTSD
* Meet DSM-IV diagnostic criteria for current substance abuse or dependence
* Be able to provide informed consent to participate in the study.

Exclusion Criteria:

* Live outside of catchment area
* Suicidal
* Pending immediate incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Crisanti, Ph.D, Principal Investigator — University of New Mexico, Department of Psychiatry, Center for Rural and Community Behavioral Health
Locations (1):
- Inside Out, Española, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because of this difficult to engage population, participants were consented and baseline data collected after they were randomized to a study arm and completed their first treatment group.
Groups:
- Peer Led: number of sessions of the intervention of an evidenced based practice called "Seeking Safety" led by a Peer (6 sessions will be used to define treatment completion)
  Seeking Safety: SS is a present-focused clinical intervention designed to target trauma/PTSD and SUDs.
- Clinician Led: number of intervention groups of an evidence based practice called "Seeking Safety" led by a master's level Clinician (6 sessions will be used to define treatment completion).
  Seeking Safety: SS is a present-focused clinical intervention designed to target trauma/PTSD and SUDs.
Period: Overall Study
Arm/Group | Peer Led | Clinician Led
Started (These individuals were determined eligible, randomized to study arms and attended 1 treatment group.) | 163 (Randomized to intervention) | 166
1st Interview Completed (These individuals attended one treatment session, were consented and completed a first interview.) | 146 | 145
3-Month Follow-Up | 94 | 95
6-Month Follow-Up | 82 | 92
Completed (Defined as completing at least one follow-up interview (3 or 6 months)) | 107 | 115
Not Completed | 56 | 51
Not completed — Lost to Follow-up | 26 | 23
Not completed — Moved Away | 1 | 2
Not completed — Incarcerated | 2 | 2
Not completed — Death | 4 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Admitted to Residential Treatment | 2 | 0
Not completed — Did not start treatment | 17 | 21

BASELINE CHARACTERISTICS:
Population: The analysis population included only those who had a baseline interview
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Led | Clinician Led | Total
Number analyzed (Participants) | 146 | 145 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10) | 35 (12) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 62 | 129
  Male | 79 | 83 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 124 | 121 | 245
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 16 | 33
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 1 | 3
  White | 86 | 90 | 176
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-traumatic Stress Disorder Symptoms
Description: PTSD Symptoms will be measured by the post-traumatic symptom checklist - civilian version. Responses are summed to yield a total severity score, with the full range for total scores being 17 to 85 (higher scores mean higher severity).
Time Frame: baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Groups:
- Peer Led: Seeking Safety Intervention Led by the Peer Providers
  Seeking Safety: SS is a present-focused clinical intervention designed to target trauma/PTSD and SUDs.
- Clinician Led: Seeking Safety Intervention Led by the Clinicians
  Seeking Safety: SS is a present-focused clinical intervention designed to target trauma/PTSD and SUDs.
Arm/Group | Peer Led | Clinician Led
Number analyzed (Participants) | 146 | 145
Score on a Scale
  Baseline | 47.2 [43.3 to 51.1] | 48.2 [44.3 to 52.1]
  3-Month Follow-Up | 43.9 [39.7 to 48.1] | 44.7 [40.5 to 48.8]
Statistical Analysis 1: Comparison: Peer Led vs Clinician Led; Test type: Non-Inferiority — Based on the PCL-C if the interventions fell within 2.5 points of each other; p = 0.01, Mixed Models Analysis; Mean Difference (Net) = 0.18, 95% CI 2-sided [-3.4 to 3.8]

2. Primary Outcome: Change in Coping Skills
Description: The Coping Scale will be used to assess coping skills. The Coping Scale directly assesses the degree to which participants report using 17 specific coping skills from SS, scaled from 0 (not at all) to 5 (extremely). This scale was selected as it is the most widely used measure of coping in the SS literature. As a result we will be able to directly compare our findings to other studies. Higher scores indicate greater frequency of use of coping skills with the range of total scores being 0 to 90
Time Frame: baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Peer Led | Clinician Led
Number analyzed (Participants) | 146 | 145
Score on a Scale
  Baseline | 45.7 [41.9 to 49.4] | 46.5 [42.8 to 50.2]
  3-Month Follow-Up | 48.6 [44.5 to 52.7] | 48.3 [44.2 to 52.4]

3. Secondary Outcome: Change in Substance Use - Alcohol Use
Description: Drug and alcohol problem severity will be assessed using the drug and alcohol subscales of the Addiction Severity Index (ASI). Items assess frequency of drug and alcohol use and abuse within the past 30 days, how bothered the individual is by his/her drug or alcohol problems, and the importance of treatment. Higher composite scores indicate more severe problems. The ASI questions focus on two distinct time periods: the past 30 days and lifetime. A number of studies have confirmed the reliability and validity of the ASI.
Time Frame: baseline, 3 months
Population: Number of Participants with an Addiction Severity Index Alcohol Composite Score greater than or equal to median of 0.0111.
Measure: Number; unit: participants
Arm/Group | Peer Led | Clinician Led
Number analyzed (Participants) | 146 | 145
participants
  Baseline | 52 | 55
  3-Month Follow-Up | 28 | 36

4. Secondary Outcome: Change in Substance Use - Drug Use
Description: as for outcome 3
Time Frame: Baseline, 3-Month
Population: Frequency of participants greater than or equal to median ASI Drug Composite Score 0.1077
Measure: Number; unit: participants
Arm/Group | Peer Led | Clinician Led
Number analyzed (Participants) | 146 | 145
participants
  Baseline | 58 | 58
  3-Month Follow-up | 24 | 31

5. Other Pre Specified Outcome: Change in Overall Mental Health
Description: Overall mental health and physical health will be assessed by the subscales of the SF-36 (short form 36). The SF-36 questions measure functional health and well-being from the patient's point of view. It is a practical, reliable, and valid measure of mental and physical health that can be completed in five to 10 minutes. The SF-36 has proven useful in differentiating the health benefits produced by different treatments. The Component Summary Scores range from 0% to 100% with higher scores indicative of higher functioning
Time Frame: baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Peer Led | Clinician Led
Number analyzed (Participants) | 146 | 145
Score on a Scale
  Basline | 36.3 [33.3 to 39.3] | 35.7 [32.7 to 38.7]
  3-Month Follow-Up | 41.2 [37.8 to 44.5] | 40.2 [36.9 to 43.5]

6. Other Pre Specified Outcome: Change in Overall Physical Health
Description: Overall mental health and physical health will be assessed by the subscales of the SF-36 (short form 36). The SF-36 questions measure functional health and well-being from the patient's point of view. It is a practical, reliable, and valid measure of mental and physical health that can be completed in five to 10 minutes. The Component Summary Scores range from 0% to 100% with higher scores indicative of higher functioning
Time Frame: baseline, 3-Month
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Peer Led | Clinician Led
Number analyzed (Participants) | 146 | 145
Score on a Scale
  Baseline | 50.8 [48.6 to 52.9] | 52.7 [50.6 to 54.9]
  3-Month Follow-Up | 50.2 [47.8 to 52.5] | 51.5 [49.2 to 53.8]

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Peer Led: ## sessions of the intervention of an evidenced based practice called "Seeking Safety" led by a Peer (6 sessions will be used to define treatment completion)
  Seeking Safety: SS is a present-focused clinical intervention designed to target trauma/PTSD and SUDs.
- Clinician Led: # intervention groups of an evidence based practice called "Seeking Safety" led by a master's level Clinician (6 sessions will be used to define treatment completion).
  Seeking Safety: SS is a present-focused clinical intervention designed to target trauma/PTSD and SUDs.
Arm/Group | Peer Led | Clinician Led
All-Cause Mortality (participants affected / at risk) | 4/146 | 3/145
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/145
Other Adverse Events (participants affected / at risk) | 0/146 | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No